CLINICAL TRIAL: NCT04147780
Title: Can the Investigators Extend the Indication for Sentinel Node Biopsy in Vulvar Cancer? A Nationwide Feasibility Study From Sweden
Brief Title: Sentinel Node Extended in Squamous Cell Vulvar Cancer
Acronym: SNEX
Status: Completed | Type: Observational
Sponsor: Diana Zach (Other)
Collaborators: Sahlgrenska University Hospital (Other); University Hospital, Linkoeping (Other); Skane University Hospital (Other)
Responsible Party: Sponsor-Investigator, Diana Zach, Principal Investigator, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Other Study IDs: 2019-04647
Record Dates: First submitted 2019-10-30; First posted 2019-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Vulva Cancer; Sentinel Lymph Node
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Primary vulvar cancer, tumor ≥ 4cm: Patients with primary squamous cell vulvar cancer, unifocal tumor ≥ 4cm:
  Sentinel node biopsy additional to radical inguinofemoral lymphadenectomy
  Interventions: Procedure: Sentinel node biopsy
- Primary vulvar cancer, multifocal tumor: Patients with primary squamous cell vulvar cancer, multifocal tumor:
  Sentinel node biopsy additional to radical inguinofemoral lymphadenectomy
  Interventions: Procedure: Sentinel node biopsy
- Local recurrence after vulvar cancer, no earlier treatment: Patients with a local recurrence of a primary squamous cell vulvar cancer, earlier without treatment of the groins or solely sentinel node biopsy:
  Sentinel node biopsy additional to radical inguinofemoral lymphadenectomy
  Interventions: Procedure: Sentinel node biopsy
- Local recurrence after vulvar cancer, earlier treatment: Patients with a local recurrence of a primary squamous cell vulvar cancer, earlier treatment of the groins by lymphadenectomy and / or (chemo-)radiation:
  Sentinel node biopsy if detectable, otherwise no groin treatment
  Interventions: Procedure: Sentinel node biopsy

INTERVENTIONS:
Procedure: Sentinel node biopsy — Sentinel node biopsy, radiotracer (mandatory) and blye dye (optional). Scintigraphy.

SUMMARY:
The aim of this study is to investigate the feasibility of sentinel node biopsy in patients with squamous cell vulvar cancer, currently not regarded suitable for the sentinel node technique, i.e. patients with tumors ≥4cm, multifocal tumors or locally recurrent disease. A positive result of this pilot study might constitute the basis for a future full-scale multinational trial.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

This study is primarily a pilot and feasibility trial, aiming to evaluate if sentinel node biopsy has a satisfactory detection rate and negative predictive value in certain groups of vulvar cancer patients.

OUTLINE:

The study is planned as a prospective, multi-center cohort study in Sweden. Since 2017, the treatment of vulvar cancer patients has been accredited to four tertiary referral university hospitals in Sweden; the Sahlgrenska University hospital in Gothenburg, the Linköping University hospital, the Skåne University hospital in Lund and the Karolinska University hospital in Stockholm.

Eligible patients will undergo a sentinel node biopsy additionally to their radical inguinofemoral lymphadenectomy and detection rate and negative predictive value for the sentinel procedure will be calculated. The study will consist of four patient groups: Patients with squamous cell vulvar cancer and:

1. primary tumors ≥4cm
2. primary multifocal tumors
3. local recurrence, earlier no treatment of the groins or only sentinel node biopsy
4. local recurrence, earlier treatment of the groins with radiotherapy / inguinofemoral lymphadenectomy

It is estimated to include 20-30 patients in each study group during a time frame of about 24 months.

RESULTS:

Results are to be expected in the end of 2021.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell vulvar cancer and

  1. primary tumors ≥ 4cm
  2. multifocal primary tumors
  3. local recurrence, earlier no treatment of the groins or only sentinel node biopsy
  4. local recurrence, earlier treatment of the groins with radiotherapy / inguinofemoral lymphadenectomy
* ≥ 18 years of age
* Considered clinically appropriate for surgery
* Informed consent

Exclusion Criteria:

* Eastern Cooperative Oncology Group performance status > 2
* Disability to read or write in Swedish
* Dementia / severe psychiatric illness leading to disability to understand the study / study information
* Signs of inguinal lymph node or distant metastases
* Ongoing pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with primary squamous vulvar cancer with tumors ≥ 4cm or multifocal tumors, and all patients with a local recurrence after primary squamous vulvar cancer in Sweden, diagnosed during the recruitment period
Sampling Method: Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2019-12-14 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Detection rate and negative predictive value for sentinel node biopsy | 2019-2021
  Calculated for each group separately. Per groin and per patient.

SECONDARY OUTCOMES:
Number of retrieved sentinel lymph nodes | 2019-2021
  Per groin
Proportion of micrometastases and isolated tumor cells, diagnosed by ultra-staging in relation to routine-histopathological examination | 2019-2021
  Per groin and per patient

CONTACTS AND LOCATIONS:
Overall Officials: Diana Zach, MD, Principal Investigator — Karolinska University Hospital, Karolinska Institute, Stockholm, Sweden
Locations (4):
- Sweden (4):
  - Karolinska University Hospital, Stockholm, Stockholm County
  - Sahlgrenska University Hospital, Gothenburg
  - Linkopings University Hospital, Linköping
  - Skanes University Hospital Lund, Lund

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Data excess requests will be reviewed by an external independent review panel. Requestors will be required to sign a data access agreement.

REFERENCES:
- [Derived] Zach D, Stenstrom Bohlin K, Kannisto P, Moberg L, Kjolhede P. Time to extend the indication for sentinel node biopsy in vulvar cancer? Results from a prospective nationwide Swedish study. Int J Gynecol Cancer. 2023 Dec 4;33(12):1845-1852. doi: 10.1136/ijgc-2023-004790. PMID 37918956
- [Derived] Zach D, Kannisto P, Stenstrom Bohlin K, Moberg L, Kjolhede P. Can we extend the indication for sentinel node biopsy in vulvar cancer? A nationwide feasibility study from Sweden. Int J Gynecol Cancer. 2020 Mar;30(3):402-405. doi: 10.1136/ijgc-2019-000938. Epub 2019 Dec 2. PMID 31796533